CLINICAL TRIAL: NCT03822104
Title: Bovine Colostrum to Fortify Human Milk for Preterm Infants: A Randomized, Controlled Trial
Brief Title: Bovine Colostrum as a Human Milk Fortifier for Preterm Infants
Acronym: FortiColos-Ⅱ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Torp Sangild (Other)
Responsible Party: Sponsor-Investigator, Per Torp Sangild, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FortiColos-CN
Record Dates: First submitted 2019-01-17; First posted 2019-01-30 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Feeding Intolerance; Necrotizing Enterocolitis; Postnatal Growth; Late-Onset Neonatal Sepsis
Keywords: Very Preterm Infants; Human Milk Fortifier; Bovine Colostrum; Enteral Feeding; Nutrition; Human milk
MeSH Terms: conditions — Enterocolitis, Necrotizing; Neonatal Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine Colostrum / intervention group (Experimental): Preterm infants are supplemented with bovine colostrum (BC) as a fortifier to human milk. BC is the first milk from cows after parturition and is a rich source of protein (80-150 g/L) and bioactive components, including lactoferrin, lysozyme, lactoperoxidase, immunoglobulins, and growth factors. The product is supplied in a sterile, powdered form and consists of unmodified, intact BC.
  Interventions: Dietary Supplement: Bovine Colostrum
- FM85 / control group (Active Comparator): Preterm infants are supplemented with PreNAN FM85 as fortifier to human milk. PreNAN FM85 contains partially hydrolyzed protein and maltodextrin including vitamins and minerals. The product is supplied in a powdered form.
  Interventions: Dietary Supplement: FM85

INTERVENTIONS:
Dietary Supplement: Bovine Colostrum — Infants randomized to the intervention group will receive a maximum of 2.8 g bovine colostrum (BC, Biofiber, Gesten, Denmark), as the HMF added to 100 ml of MM and/or DM, when EN has reached a dose of 80-100 ml/kg/d. The infants start with 1 g (0.5 g protein) BC per 100 ml human milk on the first day, increased to 2 g (1.0 g protein) on day 3, and finally 2.8 g (1.4 g protein) on day 5 if the infants only receive DM. The intervention lasts until the infants reach postmenstrual age (PMA) 35+6 weeks or in no-need of fortification due to sufficient growth, whichever comes first.
  Arms: Bovine Colostrum / intervention group
Dietary Supplement: FM85 — Infants randomized to the control group will receive a maximum of 4 g PreNAN FM85 (Nestlé, Vevey, Switzerland) as HMF, added to 100 ml MM and/or DM, when EN has reached a dose of 80-100 ml/kg/d. The infants starts with 1 g (0.35 g protein) FM85 per 100 ml human milk on the first day, which will be increased to 3 g (1.05 g protein) on day 3 and finally 4 g (1.4 g protein) on day 5, if the infants only receive DM. The infants will receive FM85 as the HMF as long as additional protein in the milk is needed until discharge.
  Arms: FM85 / control group

SUMMARY:
Very preterm infants (<32 weeks gestation) show the immaturity of organs and have high nutrient requirements for growth and development. In the first weeks, they have difficulties tolerating enteral nutrition (EN) and are often given supplemental parenteral nutrition (PN). A fast transition to full EN is important to improve gut maturation and reduce the high risk of late-onset sepsis (LOS), related to their immature immunity in gut and blood. Conversely, too fast increase of EN predisposes to feeding intolerance and necrotizing enterocolitis (NEC). Further, human milk feeding is not sufficient to support nutrient requirements for growth of very preterm infants. Thus, it remains a difficult task to optimize EN transition, achieve adequate nutrient intake and growth, and minimize NEC and LOS in the postnatal period of very preterm infants. Mother´s own milk (MM) is considered the best source of EN for very preterm infants and pasteurized human donor milk (DM) is the second choice if MM is absent or not sufficient. The recommended protein intake is 4-4.5 g/kg/d for very low birth infants when the target is a postnatal growth similar to intrauterine growth rates. This amount of protein cannot be met by feeding only MM or DM. Thus, it is common practice to enrich human milk with human milk fortifiers (HMFs, based on ingredients used in infant formulas) to increase growth, bone mineralization and neurodevelopment, starting from 7-14 d after birth and 80-160 ml/kg feeding volume per day. Bovine colostrum (BC) is the first milk from cows after parturition and is rich in protein (80-150 g/L) and bioactive components. These components may improve gut maturation, NEC protection, and nutrient assimilation, even across species. Studies in preterm pigs show that feeding BC alone, or DM fortified with BC, improves growth, gut maturation, and NEC resistance during the first 1-2 weeks, relative to DM, or DM fortified with conventional HMFs. On this background, the investigators hypothesize that BC, used as a fortifier for MM or DM, can reduce feeding intolerance than conventional fortifiers.

DETAILED DESCRIPTION:
Objectives

1. To test if fortification of human milk with BC reduces feeding intolerance compared with currently used HMF.
2. To verify the safety and tolerability of BC fortification and to monitor the rates of growth, NEC and sepsis, as investigated in a parallel trial in Denmark

Trial design This study is a dual-center, non-blinded, two-armed, randomized, controlled trial.

Participants Parents to eligible very preterm infants admitted to the Neonatal Intensive Care Units (NICU) at Nanshan People's Hospital (NAN) and Baoan Maternal and Children's Hospital in Shenzhen, China will be asked for participation.

Sample size 68 infants per group, 136 in total

Data type Clinical data

A parallel trial on BC used as human milk fortifier is conducting in Denmark (NCT03537365)

ELIGIBILITY:
Inclusion Criteria:

1. Very preterm infants born between gestational age 26 + 0 and 30 + 6 weeks (from the first day of the mother's last menstrual period and/or based on fetal ultrasound)
2. DM is given at the unit when MM is absent (or insufficient in amount)
3. Infants judged by the attending physician to be in need of nutrient fortification, as added in the form of HMF to MM and/or DM
4. Signed parental consent

Exclusion Criteria:

1. Major congenital anomalies and birth defects
2. Infants who have had gastrointestinal surgery prior to randomization
3. Infants who have received IF prior to randomization

Ages: 5 Days to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of feeding intolerance | From start of intervention until the infants reach PMA 35+6 weeks or are not in need of fortification due to sufficient growth, whichever comes first
  Number of infants in each group diagnosed with feeding intolerance for at least once. Feeding intolerance is defined as any pause of fortification or withhold of enteral feeding.

SECONDARY OUTCOMES:
Body weight | Measured weekly from the start of intervention until hospital discharge, or up to 14 weeks
  Weight gain in grams per kg body weight from birth to discharge. Weight at different time points will be calculated into z-scores according to a reference. Delta z-scores will be used to evaluate growth and for comparison between groups.
Body length | Measured weekly from the start of intervention until hospital discharge, or up to 14 weeks
  Recorded as a measure of growth in cm by standardized measuring procedures
Head circumference | Measured weekly from the start of intervention until hospital discharge, or up to 14 weeks
  Recorded as a measure of head growth in cm by standardized measuring procedures
Incidence of necrotizing entercolitis (NEC) | From the start of intervention to hospital discharge, or up to 14 weeks
  Number of infants in each group diagnosed with necrotizing enterocolitis (NEC) defined as Bell's stage II or above (Kliegman & Walsh 1987)
Incidence of late-onset sepsis (LOS) | From the start of intervention to hospital discharge, or up to 14 weeks
  Number of infants in each group diagnosed with late-onset sepsis defined as clinical signs of infection >2 days after birth with antibiotic treatment for ≥5 days (or shorter than 5 days if the participant died) with or without one positive bacterial culture in blood or cerebral spinal fluid (CSF)
Time to reach full enteral feeding | From birth to hospital discharge, or up to 14 weeks
  Number of days to full enteral feeding is reached - defined as the time when >150 ml/kg/d is reached and parenteral nutrition has been discontinued
Days on parenteral nutrition | From birth to hospital discharge, or up to 14 weeks
  Number of days that the infant receives intravenous intakes of protein and/or lipid and/or glucose
Length of hospital stay | From birth to hospital discharge, or up to 14 weeks
  Number of days in hospital, defined as days from birth until final discharge

OTHER OUTCOMES:
Volume of gastric residual | From birth to hospital discharge, or up to 14 weeks
  Volume of aspirated gastric residuals in ml
Color of gastric residual | From birth to hospital discharge, or up to 14 weeks
  The color of aspirated gastric residuals categorized into 7 colours
Incidence of bloody gastric residual | From birth to hospital discharge, or up to 14 weeks
  Number of infants in each group have had blood in the gastric residual
Frequency of stool per day | From birth to hospital discharge, or up to 14 weeks
  Frequency of stool passed each day
Amount of the stool | From birth to hospital discharge, or up to 14 weeks
  Using a 4-level pre-defined scale Amount of stool on the diaper: the percentage of area covered by stool on the diaper.
  * 1 smear;
  * 2 up to 25%;
  * 3 25-50%;
  * 4 >50%
Color of the stool | From birth to hospital discharge, or up to 14 weeks
  The color of stools categorized into 6 colors
Consistency of the stool | From birth to hospital discharge, or up to 14 weeks
  Using a 4-level pre-defined scale
Total daily volume of enteral nutrition (EN) and parenteral nutrition (PN) | From birth to hospital discharge, or up to 14 weeks
  Volume of EN (including MM, DM, infant formula, and fortification) and PN in take
Levels of macronutrients intake from EN and PN | From birth to hospital discharge, or up to 14 weeks
  Calculated based on the volume and composition of EN and PN

CONTACTS AND LOCATIONS:
Overall Officials: Per T Sangild, Study Chair — Rigshospitalet, Denmark; Ping Zhou, Principal Investigator — Shenzheng Baoan Maternity and Child Healthcare Hospital
Locations (2):
- China (2):
  - Shenzheng Baoan Maternity and Child Healthcare Hospital (SBMCH), Shenzhen, Guangdong
  - Shenzhen Nanshan People's Hospital, Shenzhen